CLINICAL TRIAL: NCT04567498
Title: eNose-TB: Electronic Nose for Tuberculosis Screening in Indonesia
Brief Title: eNose-TB: Electronic Nose for Tuberculosis Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Antonia Morita Iswari Saktiawati, Lecturer, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 002/2019
Record Dates: First submitted 2020-09-10; First posted 2020-09-28 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis
Keywords: electronic-nose; breath test; tuberculosis; screening; gender; remote area
MeSH Terms: conditions — Tuberculosis; Coitus

STUDY DESIGN:
Intervention Model Description: The Validation phase involves presumptive TB patients (Group 1) and the Screening phase involves residents of area with high risk of TB (Group 2)
Masking Description: The research subjects, breath sample takers, and laboratory sample examiners do not know the results of each sampling that has been done. The final data processor is also blinded to the results of Xpert or other laboratory examinations. The breath sampling data is saved in graphic form which interpretation will be carried out later by the data processor at the final stage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Presumptive TB patients and residents of area with high risk of TB (Experimental): Presumptive TB patients consists of 395 participants - adult and children, while Residents of area with high risk of TB consists of 1383 participants - adult and children)
  Interventions: Other: exhaled breath sampling

INTERVENTIONS:
Other: exhaled breath sampling — The participants are requested to quietly sit and breathe to the air collecting bag until the collecting bag is full. The collecting bag is sealed and connected to the e-nose machine via a collecting hose and HEPA-filter. The data are read and stored in the e-nose machine.

SUMMARY:
An electronic-nose (e-nose) is being investigated as a diagnostic tool for tuberculosis by examining exhaled breath of the patients. Universitas Gadjah Mada has developed an e-nose device for TB diagnostic tool. Here the investigators test the device in order to analyze the sensitivity and specificity electronic-nose as a screening tool for tuberculosis particularly in remote area. Various factors (gender, age, race, and location) are considered in the algorithm training to develop an inclusive eNose. Access barriers, especially those faced by women, are also assessed.

DETAILED DESCRIPTION:
The study population consists of 2 groups:

Group 1 - presumptive TB patients. Group 2 - residents of area with high risk of TB.

Study participants provide written informed consent. The participants are asked to breathe normally using a mask for 2 times then inhale and exhale in a forced expiratory volume to the air collecting bag until the collecting bag is full (two times). The collecting bag is sealed and connected to the e-nose machine via a collecting hose and HEPA-filter protecting the e-nose from microbes. The breath pattern will be recorded in the e-nose device, which is connected to a laptop that will display the recorded breath pattern. Other data are collected: clinical symptoms, results of chest X-ray, smear microscopic, and Xpert MTB/Rif examinations.

Demographic (gender, age, race, and location) and clinical data (symptoms, physical examination, laboratory examinations) are collected. Access barriers, especially for women, are also assessed through questionnaire and interviews.

ELIGIBILITY:
- Inclusion Criteria:

Validation Phase (Group 1):

* Adult and children
* Suspected of having TB
* Agree to participate in the study
* Able to produce exhaled air samples
* Able to produce samples for Xpert MTB/Rif examination

Screening Phase (Group 2):

* Adult and children
* Agree to participate in the study
* Able to produce exhaled air samples
* Currently not in TB treatment

  - Exclusion Criteria
* Invalid measurements of breath tests
* Incomplete CXR data
* Missing specimens
* Unable to breath normally for 2 minutes due to respiratory illness

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1778 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of electronic nose signal in screening tuberculosis that is measured through sensitivity, specificity, PPV, NPV | 2 years
  sensitivity, specificity, positive predictive value, negative predictive value of e-nose signal in diagnosing TB, factors influencing the diagnostic accuracy
Access barriers, measured through questionnaire, interview, and focus group discussion | 2 years
  access barriers to the TB screening that are measured through questionnaire, interview, and focus group discussion

SECONDARY OUTCOMES:
Time of a screening algorithm with eNose-TB, measured in days | 2 years
  Time of a screening algorithm with eNose-TB to obtain additional detection of one TB case, measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Saktiawati, MD, PhD, Principal Investigator — Faculty of Medicine, Public Health and Nursing Universitas Gadjah Mada
Locations (3):
- Indonesia (3):
  - Balai Kesehatan Masyarakat Klaten, Klaten, Central Java
  - Primary health centers and hospital, Timika, Special Region of Papua
  - Primary health centers and hospital, Yogyakarta, Special Region of Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saktiawati AMI, Triyana K, Wahyuningtias SD, Dwihardiani B, Julian T, Hidayat SN, Ahmad RA, Probandari A, Mahendradhata Y. eNose-TB: A trial study protocol of electronic nose for tuberculosis screening in Indonesia. PLoS One. 2021 Apr 21;16(4):e0249689. doi: 10.1371/journal.pone.0249689. eCollection 2021. PMID 33882070